CLINICAL TRIAL: NCT03283124
Title: A Multicenter Randomized Controlled Non-inferiority Trial Comparing Transvaginal Self-tailored Titanium-coated Polypropylene Mesh Procedure With Mesh-kit Procedure.
Brief Title: Comparing Transvaginal Self-tailored Titanium-coated Polypropylene Mesh Procedure With Mesh-kit Procedure.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Collaborators: Shanghai Medstron Medical Co.Ltd (Unknown); LinkDoc Technology (Beijing) Co. Ltd. (Industry); Chinese Academy of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: self-cut mesh vs mesh-kit
Record Dates: First submitted 2017-05-07; First posted 2017-09-14 (Actual); Last update posted 2019-03-05 (Actual); Status verified 2019-02

CONDITIONS: Pelvic Organ Prolapse
MeSH Terms: conditions — Pelvic Organ Prolapse

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: participant and investigator are not blinded. outcome assessor who are in charge of follow-up assement is masked.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- self-cut mesh procedure (Active Comparator): This procedure is transvaginal mesh implantation surgery for POP patients. Self-cut mesh procedure is an economic pelvic reconstructive surgical operation with use of specially designed puncture needles and self-cut mesh, which mainly provide anterior and apical compartments support, with posterior compartment reinforced by bridge technique repair. The mesh pieces used in this surgery was cut from a single piece of mesh material(TiLOOP 10*15cm) which is much cheaper and readily available. Patients could have transvaginal hysterectomy concomitantly.
  Interventions: Procedure: pelvic floor reconstructive surgery
- mesh-kit procedure (Active Comparator): This procedure is transvaginal mesh implantation surgery for POP patients.Mesh-kit procedure is refered to pelvic floor reconstructive surgery with titanium-coated meshes kit(TiLOOP TOTAL6).Patients could have transvaginal hysterectomy concomitantly.
  Interventions: Procedure: pelvic floor reconstructive surgery

INTERVENTIONS:
Procedure: pelvic floor reconstructive surgery — transvaginal mesh implantation for pelvic organ prolapse

SUMMARY:
Pelvic organ prolapse(POP) is a common health problem and has significant negative effects on woman's quality of life. Transvaginal mesh procedure is a durable reconstructive surgery, but the mesh kits are expensive for underdeveloped countries. Our preliminary trial showed that the use of self-tailored mesh had good success rate (91.8% at 1-year follow-up) and low complication rate. The trial is designed to compare self-tailored titanium-coated polypropylene mesh procedure with mesh-kit in the treatment of POP stage III-IV in terms of efficacy, safety and cost-effective .

DETAILED DESCRIPTION:
The trial is a randomized controlled multi-center non-inferiority trial. The primary outcome measure is success rate at 1-year follow-up. The second outcomes are subjective improvement of quality of life, complications and costs. Analysis will be performed according to the intention to treat principle. Based on comparable success rate of 90% and 10% as the margin(beta 0.2 and one sided alpha 0.025), about 312 patients in total from 11 centers will be recruited per group including 10% drop-out. The aims of the research are to demonstrate whether self-tailored mesh is non-inferior to the mesh-kit. The finding of this research might influence the treatment selection for POP in China.

ELIGIBILITY:
Inclusion Criteria:

* Age:More than 50 years old with 3 years after menopause or more than 55 years old, but less than 75 years old.
* Subject must have severe apical or anterior vaginal prolapse (stage III-IV), with moderate posterior vaginal prolapse(stage I-II). This is defined as ( C > +1cm OR Ba > +1cm, with Bp ≤+1cm by the POP-Q). This is the most common modality of multiple compartment POP in clinic.
* Subject reports a bothersome bulge they can see or feel per PFDI-20, question 3, response of 2 or higher (i.e., responses of "somewhat", "moderately", or "quite a bit").
* Desires transvaginal mesh treatment for primary or recurrent, symptomatic uterovaginal prolapse.
* Concomitant hysterectomy when indicated. But concomitant anti-incontinence surgeries will not be enrolled.
* Subject is willing and able to comply with the follow-up regimen.

Exclusion Criteria:

* Subject is pregnant or intends to become pregnant in the future
* Subject has an active or chronic systemic infection including any gynecologic infection, untreated urinary tract infection (UTI) or tissue necrosis
* Subject has history of pelvic organ cancer (e.g. uterine, ovarian, bladder, colo-rectal or cervical)
* Subject has had prior or is currently undergoing radiation, laser therapy, or chemotherapy in the pelvic area
* Subject has taken systemic steroids (within the last month), or immunosuppressive or immunomodulatory treatment (within the last 3 months)
* Subject has systemic connective tissue disease (e.g. scleroderma, systemic lupus erythematosus (SLE), Marfan syndrome, Ehlers Danlos, collagenosis, polymyositis, polymyalgia rheumatica)
* Subject has chronic systemic pain that includes the pelvic area or chronic focal pain that involves the pelvis
* Subject has uncontrolled diabetes mellitus (DM)
* Subject has a known neurologic or medical condition affecting bladder function (e.g., multiple sclerosis, spinal cord injury or stroke with residual neurologic deficit)
* Subject has had previous prolapse repair with mesh in the target compartment

Ages: 50 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 312 (Estimated)
Dates: Start 2018-01-12 (Actual); Primary Completion 2020-01-12 (Estimated); Study Completion 2022-01-12 (Estimated)

PRIMARY OUTCOMES:
surgical "success" | up to 36 months after operation
  Subjects will be considered a success if they meet the definitions of anatomic cure and deny vaginal bulging symptoms, and no additional treatment for prolapse(surgical or pessary use).
  Anatomic cure is defined as leading edge above the hymen (i.e Ba, C, Bp<0 cm) Symptomatic cure is defined as the absence of vaginal bulge symptoms as indicated by a negative response question 3 of the pelvic floor distress inventory- 20 (PFDI-20): "Do you usually have a bulge or something falling out that you can see or feel in your vaginal area?

SECONDARY OUTCOMES:
anatomic outcomes | up to 36 months after operation
  anatomic outcome of each vaginal segment( anterior, posterior and apical) using POP-Q score.
symptomatic improvement using validated instruments(PFIQ-7) | up to 36 months after operation
  Relief of symptoms using validated instruments(PFIQ-7) .
symptomatic improvement using validated instruments(PFDI-20) | up to 36 months after operation
  Relief of symptoms using validated instruments(PFDI-20) .
symptomatic improvement using validated instruments(PISQ-12) | up to 36 months after operation
  Relief of symptoms using validated instruments(PISQ-12)
symptomatic improvement using patient global impression of change (PGI-C) | up to 36 months after operation
  Relief of symptoms using patient global impression of change (PGI-C)
intraoperative and post operative complications | up to 36 months after operation
  using IUGA/ICS joint terminology CTS coding system and dingo system
post operative pain | within 3 days after operation
  visual analogue scales (VAS) were used to evaluate the degree of pain.
Hospital costs | up to 4 weeks after operation
  hospitlization expenses

CONTACTS AND LOCATIONS:
Overall Officials: Lan Zhu, Principal Investigator — Peking Union Medical College Hospital
Locations (11):
- China (11):
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - Fosha Maternal and Child Health Care Hospital, Foshan, Guangdong
  - The First Affiliated Hospital of Guangzhou Medical College, Guangzhou, Guangdong
  - Changsha Maternal and Child Health Care Hospital, Changsha, Hunan
  - The second Xiangya Hospital of Central South University, Changsha, Hunan
  - Wuxi Maternal and Child Health Care Hospital, Wuxi, Jiangsu
  - Qilu Hospital of Shandong University, Jinan, Shandong
  - Shanxi Provincial People's Hospital, Xi’an, Shanxi
  - Sichuan University West China Second University Hospital, Chengdu, Sichuan
  - the First Affiliated Hospital of Xinjiang Medical University, Ürümqi, Xinjiang
  - the People's Hospital of Xinjiang Uygur Autonomous Region, Ürümqi, Xinjiang

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chen J, Yu J, Morse A, Tao G, Gong J, Wang B, Wang Y, Ababaikeli G, Jiang X, Liu P, Zhang X, Nisier H, Wang P, Funfgeld C, Huang K, Zhang H, Sun X, Zhu L. Effectiveness of Self-cut vs Mesh-Kit Titanium-Coated Polypropylene Mesh for Transvaginal Treatment of Severe Pelvic Organ Prolapse: A Multicenter Randomized Noninferiority Clinical Trial. JAMA Netw Open. 2022 Sep 1;5(9):e2231869. doi: 10.1001/jamanetworkopen.2022.31869. PMID 36112377
- [Derived] Chen J, Yu J, Morse A, Funfgeld C, Huang K, Gong J, Tao G, Wang B, Wang Y, Jiang X, Ababaikeli G, Liu P, Nisier H, Zhang X, Wang P, Sun X, Zhu L. Self-cut titanium-coated polypropylene mesh versus pre-cut mesh-kit for transvaginal treatment of severe pelvic organ prolapse: study protocol for a multicenter non-inferiority trial. Trials. 2020 Feb 26;21(1):226. doi: 10.1186/s13063-019-3966-3. PMID 32102687